CLINICAL TRIAL: NCT06995573
Title: A Phase 2a, Multi-Center, Randomized, Parallel Group, Double Blind and Placebo-controlled Clinical Trial to Assess Safety and Tolerability as Well as Explorative Efficacy of the Orthosteric Selective Muscarinic M1 Agonist NSC001 in Mild to Moderate Alzheimer's Disease
Brief Title: A Study to Assess Safety and Tolerability and to Explore Efficacy of NSC001 in Mild to Moderate Alzheimer's Disease
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NSC-Therapeutics (Industry)
Collaborators: NeuroScios GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NSC24001; 2024-518563-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-04-02; First posted 2025-05-29 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
Keywords: Mild to Moderate Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): 40 mg QD of NSC001
  Interventions: Drug: NSC001
- Arm 2 (Experimental): 40 mg QD of NSC001 + 20 mg of Trospium
  Interventions: Drug: NSC001
- Arm 3 (Placebo Comparator): Placebo: with or without 20 mg of Trospium
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NSC001 — rigid, orthosteric acetylcholine analog, highly specific for M1 muscarinic receptor
  Arms: Arm 1; Arm 2
Other: Placebo — matching placebo to NSC001
  Arms: Arm 3

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of NSC001 on in patients with mild to moderate Alzheimer's disease and to evaluate the influence of the compound on cognitive function.

DETAILED DESCRIPTION:
NSC001 is an orally administered small molecule rigid cholinergic agonist that has a high selectivity for M1 muscarinic receptors (MI), designed to improve cognitive and behavioral function in patients with Alzheimer's Disease (AD). The primary pharmacology available for NSC001 from preclinical models and studies in healthy volunteers provides a compelling rationale for the evaluation of the safety and tolerability of this compound in patients with mild to moderate AD and for the investigation of NSC001 effects on cognitive function and behavior in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants and competent trial partner/caregiver are willing and able to give signed informed consent for participation in the trial including compliance with the requirements and restrictions according to local regulations for the trial Informed Consent Form (ICF). Signed informed consent by the patient (examined and verified to be mentally capable by an independent physician/ neurologist) prior to the initiation of any study specific procedure.
* Must have an informant or trial partner who, in the Investigator's judgment, has frequent and sufficient contact with the participant (at least 10 hours/week), who is considered reliable by the Investigator in providing support to the participant to ensure compliance with the trial intervention, including the proper and consistent intake of the study medication, who can accompany the participant to trial visits and help with protocol procedures, and who is also able and willing to provide input for completing the caregiver scales and sign the caregiver consent form.
* Male or female aged 50 to 85 years, inclusive at the time of consent.
* Female trial participants must be post-menopausal for at least 2 consecutive years or surgically sterile (bilateral tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 6 months prior to screening.
* Male trial participants with partners who are women of childbearing potential (WOCBP) must agree to use a reliable means of contraception (e.g., minimum condom + spermicide) during the trial and 6 months after discontinuing the trial intervention
* Participants who have a clinical diagnosis of AD, which falls into the stages of mild to moderate dementia (Stage 4 to 5) according to the utilized by the NIA-AA 2018 criteria at screening.
* Patients who show CSF biomarker data supporting the diagnosis of AD measured within the last 3 years or patients with a positive Amyloid Pet Scan within the last 3 years or have a test on p-tau217 in plasma indicating brain amyloid positivity will qualify for the study. Plasma pTau217 concentration of ≥ 2.0 pg/mL.
* Evidence of cognitive decline over the last year must be present based on informant observation, medical records, or objective neurocognitive testing.
* Magnetic resonance imaging (MRI) or computed tomography (CT) scan performed within 12 months before screening, with findings consistent with the clinical diagnosis of mild to moderate AD without any other clinically significant comorbid pathologies, especially cerebrovascular lesions. If an MRI or CT scan is unavailable within 12 months before screening, an MRI assessment should be completed, and the findings confirmed before the participant's treatment start (V1).
* Mini-Mental State Examination (MMSE) score of ≥18 and ≤26 at screening.
* Modified Hachinski Ischemic (mHIS) Scale ≤4 unless recent MRI study demonstrates no vascular causes for dementia.
* Use of AChEIs (e.g., donepezil, galantamine, or rivastigmine) is mandatory and treatment must be on a stable dose for at least 3 months prior to baseline
* Adequate vision, hearing, and motor function to comply with testing.
* Ability to swallow size 2 capsules.
* In the opinion of the Investigator is in reasonably good health for 21-week trial participation.
* Trial participants must consent to ApoE genotyping. Their ApoE status may be disclosed to the participant at the Investigator's discretion.

Exclusion Criteria:

* Inability to comply with visit schedule or other protocol requirements and failure to perform screening and baseline first treatment visit (V1) assessments.
* Planned start of NMDA receptor antagonist memantine during the trial period (i.e., the next 13 weeks) or use of memantine within the past 4 weeks before screening, unless at a stable dose for at least 8 weeks prior to screening.
* Prior use of anti-beta-amyloid immunotherapy (e.g., Aducanumab, Leqanemab, Donanemab) or administration of anti-amyloid vaccine.
* Enrollment in another investigational clinical trial and, respectively, administration of investigational drug within the previous 3 months small molecules. Previous participation in investigational clinical trials with monoclonal antibodies against amyloid or other anti-beta amyloid immunotherapy and other biologicals.
* Current use of anticholinergics, including trospium within the past 2 weeks before screening.
* Use of the following medications:

  1. Long-acting benzodiazepines (e.g., valium), except for sedation prior to screening MRI scans for those participants requiring sedation and should not be administered within 24 hours prior to cognitive testing.
  2. Short/medium-acting benzodiazepines (e.g., alprazolam, lorazepam, oxazepam, temazepam) except if used chronically for sleep and on a stable dose for ≥4 weeks prior to screening and throughout the trial. May not be taken within 12 hours prior to cognitive testing.
  3. Sedating antihistamines if taken within 12 hours prior to cognitive testing (Non-sedating antihistamines [e.g., fexofenadine, cetirizine] are allowed).
  4. Anticonvulsants that have significant effects on cognition per the Investigator's opinion and/or anticonvulsants used for treatment of seizures. Anticonvulsants with limited cognitive effects, such as lamotrigine, pregabalin, levetiracetam for the treatment of pain, and other non-epilepsy indications are allowed if, in the opinion of the Investigator, they are not producing sedation or contributing to cognitive impairment. The participant must have been on a stable dose for ≥4 weeks prior to screening and throughout the trial.
  5. Antidepressants that may, in the Investigator's opinion, affect the participant's cognition (e.g., tricyclic antidepressants). Mild depression or depressive mood arising in the context of AD are not criteria for exclusion. Use of antidepressants is allowed if at stable doses for ≥4 weeks prior to screening and throughout the trial.
  6. Antipsychotics used regularly, except for low doses of atypical antipsychotics (e.g., risperidone, aripiprazole, or quetiapine) if used on an as-needed basis or if used at a stable dose for ≥4 weeks prior to screening and throughout the duration of the trial. The definition of "low doses" should be judged by the Investigator, and the Medical Monitor can be consulted if needed.
  7. Prior use of levodopa or anti-Parkinsonian medications including dopaminergic agents, amantadine, selegiline, benztropine, and monoamine oxidase (MAO) inhibitors prescribed for the treatment of Parkinsonism or Parkinson's disease.
  8. Use of prescription narcotic medications within 4 weeks prior to screening. After randomization, short-term use of prescription narcotics is allowed for specific situations (e.g., after surgical procedures) and if administered at least 24 hours prior to cognitive testing.
  9. Use of drugs with known QT-prolonging effects36, unless used at a stable dose for ≥12 weeks prior to screening and throughout the duration of the trial, and with demonstrated stable QT interval on treatment.
  10. Use of any drug of abuse, including but not limited to, amphetamine, cannabis, cocaine, opiate, propoxyphene, methadone, methaqualone, phencyclidine, or barbiturates.
  11. Centrally active anti-hypertensive drugs (clonidine, l-methyl DOPA, guanidine, guanfacine, etc.).
* Hospitalization or change of chronic concomitant medication within 4 weeks prior to screening or during screening period.
* Clinical, laboratory or neuro-imaging findings consistent with:

  1. Other primary degenerative dementia, (e.g., dementia with Lewy bodies, fronto temporal dementia, Parkinson's disease, Huntington's disease, Creutzfeldt-Jakob's disease, Down's syndrome, etc.).
  2. Other neurodegenerative condition (e.g., Parkinson's disease, Amyotrophic Lateral Sclerosis, etc.).
  3. Cerebrovascular disease (major infarct, 1 strategic or multiple lacunar infarcts, extensive white matter lesions >one quarter of the total white matter) based on historical or current CT or MRI.
  4. Other CNS diseases (e.g., severe head trauma, tumors, subdural hematoma, or other space-occupying processes, etc.).
  5. Seizure disorder, except history of febrile seizures in childhood.
  6. Other infectious, metabolic, or systemic diseases affecting the CNS (e.g., syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, serum electrolytes out of normal range, juvenile-onset diabetes mellitus, etc.).
* A current Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) diagnosis of active major depression, schizophrenia, or bipolar disorder or are at suicide risk, as determined by meeting any of the following criteria:

  1. Suicide attempt within the past 12 months prior to screening.
  2. Suicidal ideation as defined by a positive response to questions 4 and 5 on the C-SSRS within 60 days of screening.
* Have a history of substance abuse (based on DSM-IV criteria) within the past 12 months prior to screening, a positive urine drug (due to nonprescription drug) or alcohol test at screening, or use of cannabinoids (prescription or recreational).
* Significant acute or chronic infection at screening including, among others: History of, or positive test result at screening visit for, human immunodeficiency virus (HIV) or known current hepatitis C or hepatitis B virus infection, or positive test result at screening (defined as hepatitis B virus [HBV] surface Ag positive or positive HCV with reflex to positive hepatitis C virus [HCV] RNA).
* Clinically significant, advanced, or unstable disease that may interfere with primary or secondary variable evaluations, and which may bias the assessment of the clinical or mental status of the trial participant or put the participant at special risk, such as:

  1. Respiratory insufficiency.
  2. Heart disease (myocardial infarction, unstable angina, heart failure, cardiomyopathy within 6 months before screening).
  3. Bradycardia (heartbeat <50/min) or tachycardia (heartbeat >100/min), confirmed by repeat measurement.
  4. Higher degree AV block (Mobitz type II and III), congenital long QT syndrome, sinus node dysfunction or prolonged QTcF-interval (males >450 msec and females >470 msec).
  5. Uncontrolled hypertension (>180/95 mm Hg) or hypotension (<90/60 mm Hg or higher if symptomatic), confirmed by repeat measurement.
* Indication of impaired renal function at screening defined as creatinine clearance ≤60 mL/min according to Chronic Kidney Epidemiology Collaboration (CKD-EPI) formula (confirmed by repeat measurement).
* Indication of uncontrolled diabetes at screening defined by HbA1c >8.5%.
* Indication of chronic liver disease, liver function test abnormalities, or other signs of hepatic insufficiency (alanine transaminase [ALT], aspartate aminotransferase [AST], gamma-glutamyl transferase (GGT), or alkaline phosphatase [ALP] >2.5 upper limit of normal [ULN]; confirmed by repeat measurement).
* History of pre-malignant or malignant disease. The following exceptions may be made after discussion with the Sponsor:

  1. Participants with cancers in remission ≥5 years prior to screening.
  2. Participants with a history of excised or treated basal cell or squamous carcinoma of the skin.
  3. Participants with localized prostate cancer with treatment cycles that were completed at least 6 months prior to screening.
* Suspected or known allergy to any components of the trial interventions.
* Any condition, which, in the opinion of the Investigator, makes the trial participant unsuitable for inclusion.
* If the trial participant is in any way dependent on the Sponsor or the Investigator or if the trial participant is accommodated in an establishment on a judicial or administrative order.
* Female participants who are pregnant or currently breastfeeding or who plan to become pregnant.
* Male participants with a partner who is pregnant or currently breastfeeding or who plans to become pregnant.
* In case an MRI is needed at screening, contraindications to having a brain MRI (e.g., MRI-incompatible pacemaker, MRI-incompatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia that cannot be medically managed).
* Any contraindication to trospium chloride, including known hypersensitivity to trospium chloride or any of the excipients listed in the SmPC, myasthenia gravis, urinary retention, gastric retention, toxic megacolon, ulcerative colitis or uncontrolled narrow-angle glaucoma.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of NSC001 | Week 0 and week16
  Number of Adverse Events (AEs) between V1 (Baseline) -V5 (End of Treatment)
Safety during the treatment period | Week 0 and week16
  Number of Serious Adverse Events (SAEs) between V1 (Baseline) -V5 (End of Treatment)

SECONDARY OUTCOMES:
Maximum concentration in plasma | At week 0, 1, 2, 3, 4, 16 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4 and 6 hours)
  Maximum concentration of NSC001 in Plasma, C (max)
Time at maximum concentration in plasma | At week 0, 1, 2, 3, 4, 16 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4 and 6 hours)
  Time at maximum concentration of NSC001 in Plasma, T(max)
Area under the curve | At week 0, 1, 2, 3, 4, 16 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4 and 6 hours)
  Area under the curve; Concentration of NSC001 in blood plasma as a function of time.
Half Life of NSC001 in plasma | At week 0, 1, 2, 3, 4, 16 at pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4 and 6 hours)
  Half Life of NSC001; The time it takes for the concentration of NSC001 in the plasma to be reduced by 50%

OTHER OUTCOMES:
ADAS-cog as exploratory outcome on cognitive function and neuropsychiatric symptoms | At week 0, 4, 16
  Alzheimer's disease Assessment Scale (ADAS-Cog) The ADAS-Cog measures the cognitive decline over time. The increase of the ADAS-cog score indicates a worsening of the disease. The score goes from 0 to 85max.
MMSE as exploratory outcome on cognitive function and neuropsychiatric symptoms | At week 0, 1, 2, 3, 4, 16
  Mini Mental State Examination (MMSE) The MMSE measures the cognitive decline over time. The decrease of the MMSE score indicates a worsening of the disease. The score goes from 0 to 30max. For the study an MMSE between 18 -26 is required. Subjects with a lower or higher MMSE are excluded.
Concentration of NFL as exploratory outcome on blood-based AD-related biomarkers | At week 0,4,16
  Concentration of Neurofilament light chain (NFL) as biomarker for neuronal damage.
Concentration of Amyloid Beta (AB42) as exploratory outcome on blood-based AD-related biomarkers | At week 0,4,16
  Concentration of Amyloid Beta (AB42) as key biomarker for Alzheimer's Disease.
Concentration of Amyloid Beta (AB40) as exploratory outcome on blood-based AD-related biomarkers | At week 0,4,16
  Concentration of Amyloid Beta (AB40) as key biomarker for Alzheimer's Disease.
Tau concentration as blood-based AD-related biomarker | At week 0,4,16
  Concentration of total Tau as key biomarker for Alzheimer's Disease.
p-Tau181 concentration as blood-based AD-related biomarker | At week 0,4,16
  Concentration of p-Tau181 as key biomarker for Alzheimer's Disease.
p-Tau217 concentration as blood-based AD-related biomarker | At week 0,4,16
  Concentration of p-Tau 217 as key biomarker for Alzheimer's Disease.
Exploratory outcome on QTc interval | 16 weeks
  To evaluate the effects of NSC001, with or without trospium, on QTc interval (Fridericia correction to be used)

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Windisch, PhD, Study Chair — NSC-Therapeutics GmbH
Locations (6):
- Austria (2):
  - University Hospital Graz, Graz, Styria
  - Gemeinnuetzige Salzburger Landeskliniken Betriebsgesellschaft GmbH, Salzburg
- Germany (4):
  - Zentrum fuer klinische Forschung Dr. I. Schoell GmbH, Bad Homburg
  - Universitaetsmedizin Goettingen, Göttingen
  - Dynamikos GmbH Institut fuer Studien zur Psychischen Gesundheit, Mannheim
  - Rostock University Medical Center, Rostock

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fisher A. Cholinergic modulation of amyloid precursor protein processing with emphasis on M1 muscarinic receptor: perspectives and challenges in treatment of Alzheimer's disease. J Neurochem. 2012 Jan;120 Suppl 1:22-33. doi: 10.1111/j.1471-4159.2011.07507.x. Epub 2011 Nov 28. PMID 22122190
- [Background] Fisher A. Cholinergic treatments with emphasis on m1 muscarinic agonists as potential disease-modifying agents for Alzheimer's disease. Neurotherapeutics. 2008 Jul;5(3):433-42. doi: 10.1016/j.nurt.2008.05.002. PMID 18625455